CLINICAL TRIAL: NCT03512847
Title: Predictive Gene Profiles and Dynamic Measurement of Treatment Response in Metastatic Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REG-006-2018
Record Dates: First submitted 2018-03-26; First posted 2018-05-01 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Nonsmall Cell Lung Cancer
Keywords: liquid biopsy; genomic profiling; ctDNA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Comprehensive molecular profiling. Whole Exome Sequencing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims include:

* Exploring potential predictive molecular profiles to immunotherapy/chemotherapy
* Investigating the role of circulating tumor DNA as a dynamic biomarker during immunotherapy/chemotherapy
* Identifying possible resistance mechanisms to immunotherapy/chemotherapy

Materials and methods:

Approximately 150 patients diagnosed with metastatic NSCLC assigned for immunotherapy or chemotherapy will be candidates for inclusion during a 1-2 years period.

A comprehensive molecular profiling will be made from the diagnostic biopsy. Before every treatment-cycle a blood sample will be taken to quantify ctDNA. At time of progressive disease during/after first line treatment, patients will be asked to participate in a new biopsy and a comprehensive molecular profiling will be performed.

The tissue and blood samples collected will be stored in a biobank. Clinical data will be collected to perform a comprehensive database.

Analysis:

Potentially predictive molecular profiles for immunotherapy/chemotherapy will be found by comparison of treatment outcome for patients with specific molecular characteristics.

Through quantification of ctDNA during treatment and upon progression, the role of ctDNA as a dynamic biomarker will be further strengthened.

Differences in molecular profiles pre- and post-treatment may reveal resistance mechanisms to treatment. Molecular profiling on progression can be valuable in second-line treatment guidance.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Able to understand and read Danish
* WHO Performance status 0-2
* Acceptable organ function (liver/kidney/heart) for treatment
* The disease has to be:

evaluable or measurable according to RECIST/iRECIST accessible for biopsy metastatic or not suitable for curative intended treatment

Exclusion Criteria:

* Other active cancers
* Contraindications for systemic therapy
* ALK-positive, ROS-1 or EGFR mutations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic non-small cell lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
Predictive gene profiles | until progression or death, an average of 3 years
  Concordance between specific gene profiles and treatment outcomes
Resistance mechanisms toward chemotherapy and immunotherapy | until progression or death, an average of 3 years
  Differences in molecular profiles pre- and post-treatment
ctDNA as a dynamic biomarker | until progression or death, an average of 3 years
  Quantification of ctDNA during treatment linked to treatment outcome

CONTACTS AND LOCATIONS:
Overall Officials: Frank S Malene, MD, Principal Investigator — Region Zeland
Locations (1):
- Department of Oncology, Næstved, Region Sjælland, Denmark

REFERENCES:
- [Derived] Frank MS, Andersen CSA, Ahlborn LB, Pallisgaard N, Bodtger U, Gehl J. Circulating Tumor DNA Monitoring Reveals Molecular Progression before Radiologic Progression in a Real-life Cohort of Patients with Advanced Non-small Cell Lung Cancer. Cancer Res Commun. 2022 Oct 13;2(10):1174-1187. doi: 10.1158/2767-9764.CRC-22-0258. eCollection 2022 Oct. PMID 36969747
- [Derived] Frank MS, Bodtger U, Hoegholm A, Stamp IM, Gehl J. Re-biopsy after first line treatment in advanced NSCLC can reveal changes in PD-L1 expression. Lung Cancer. 2020 Nov;149:23-32. doi: 10.1016/j.lungcan.2020.08.020. Epub 2020 Sep 12. PMID 32949828